CLINICAL TRIAL: NCT00000122
Title: Fluorouracil Filtering Surgery Study (FFSS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NEI-21
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Fluorouracil

INTERVENTIONS:
Drug: 5-Fluorouracil

SUMMARY:
To determine whether postoperative subconjunctival injections of 5-fluorouracil (5-FU) increase the success rate of filtering surgery in patients at high risk for failure after standard glaucoma filtering surgery.

DETAILED DESCRIPTION:
Filtering surgery adequately lowers intraocular pressure in most glaucoma patients. However, the prognosis is less favorable for aphakic patients with glaucoma or glaucoma in phakic eyes following unsuccessful filtering operations. Failure of filtering surgery is usually attributed to the proliferation of fibroblasts at the filtering site. The use of 5-FU, an antimetabolite, has been shown to inhibit the proliferation of fibroblasts in tissue culture, and in preliminary studies it has increased the success of filtering surgery in a nonhuman primate model.

The Fluorouracil Filtering Surgery Study (FFSS) was a randomized, controlled clinical trial comparing the success rate of standard glaucoma filtering surgery to the success rate of standard surgery with adjunctive 5-FU treatment.

Another element of this study was to evaluate the frequency and severity of possible adverse effects related to 5-FU injections. Detailed preoperative and postoperative examinations of the cornea, lens, and retina were performed. Systemic toxicity was assessed by preoperative and postoperative hematologic studies.

After the investigators performed the filtering surgery and determined that the new outlet channel was working, patients were randomized to receive either 5-FU injections or standard postsurgical care without 5-FU. The patients treated with 5-FU received subconjunctival injections of 5 mg of 5-FU twice daily on postoperative days 1 through 7 and once daily on postoperative days 8 through 14. There were 213 patients recruited into the study, 162 with previous cataract extraction and 51 with previous filtering surgery.

All patients were examined at 1 month, 3 months, 6 months, 1 year, 18 months, and 2 years postoperatively and at yearly intervals thereafter until 5 years postoperatively. Possible concomitant risks of 5-FU treatment, such as toxic effects to the cornea, lens, or retina, were monitored.

ELIGIBILITY:
Men and women with uncontrolled intraocular pressure greater than 21 mm Hg in one or both eyes despite maximal tolerated therapy and who were aphakic or had undergone previous filtering surgery were eligible to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1985-09; Study Completion 1988-06 (Actual)

REFERENCES:
- [Background] Fluorouracil Filtering Surgery Study one-year follow-up. The Fluorouracil Filtering Surgery Study Group. Am J Ophthalmol. 1989 Dec 15;108(6):625-35. doi: 10.1016/0002-9394(89)90853-2. PMID 2688428
- [Background] Risk factors for suprachoroidal hemorrhage after filtering surgery. The Fluorouracil Filtering Surgery Study Group. Am J Ophthalmol. 1992 May 15;113(5):501-7. doi: 10.1016/s0002-9394(14)74720-8. PMID 1575223
- [Background] Three-year follow-up of the Fluorouracil Filtering Surgery Study. Am J Ophthalmol. 1993 Jan;115(1):82-92. doi: 10.1016/s0002-9394(14)73529-9. PMID 8420383
- [Background] Five-year follow-up of the Fluorouracil Filtering Surgery Study. The Fluorouracil Filtering Surgery Study Group. Am J Ophthalmol. 1996 Apr;121(4):349-66. doi: 10.1016/s0002-9394(14)70431-3. PMID 8604728